CLINICAL TRIAL: NCT00243568
Title: Vicriviroc (SCH 417690) in Combination Treatment With Optimized ART Regimen in Experienced Subjects (VICTOR-E2)
Brief Title: Vicriviroc, a CCR5 Inhibitor, Added to an Optimized Antiretroviral Therapy for Previously Treated HIV (VICTOR-E2) (Study P04285
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04285; EudraCT number 2005-001058-26
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; CCR5/CXCR4 mixed tropism; R5/X4 mixed tropism; CCR5 inhibitor; vicriviroc; treatment-experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vicriviroc

INTERVENTIONS:
Drug: Vicriviroc

SUMMARY:
This is an international study of vicriviroc in 500 adult HIV-infected subjects who are failing standard antiretroviral therapy (ART). HIV must be of a certain type known as R5/X4-mixed tropic. Subjects allowed into the trial will be randomly assigned to treatment with vicriviroc 10 mg QD, vicriviroc 15 mg QD, or placebo in addition to other antiretrovirals (selected by the investigator to be optimal for the specific subject) containing at least 3 drugs, including a protease inhibitor (PI) boosted with at least 100 mg ritonavir QD. Subjects will be continued for up to 48 weeks of dosing.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, multi-site, parallel-group, double-blind study of vicriviroc (SCH 417690) in 500 adult HIV-infected subjects with R5/X4 mixed viral tropism who have at least 5000 copies/mL HIV RNA despite standard antiretroviral therapy (ART) that the subject has been receiving continuously for at least 3 months. Eligible subjects will be randomized to treatment with vicriviroc 10 mg QD, vicriviroc 15 mg QD, or placebo in addition to an individually optimized PI-containing ART regimen containing at least 3 drugs, including a PI, boosted by at least 100 mg ritonavir QD prescribed by the investigator. The vicriviroc dose and placebo will be double-blind, and the optimized background therapy will be open-label. Treatment visits after Day 1 are scheduled for Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48. A planned interim analysis will be conducted when 100 subjects have completed 12 weeks of dosing. After completion of the primary analysis (24-week virologic response of all subjects), subjects will be given the optimal dose of vicriviroc and follow-up will be continued to at least 48 weeks. Safety will be monitored by standard laboratory tests, assessment of adverse events, and emergence of complicating medical conditions. Cardiac safety will be monitored periodically by ECG, and plasma samples will be collected from all subjects through the study for population pharmacokinetic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with documented R5/X4 mixed-tropic HIV infection
* Prior therapy for greater than or equal to 3 months with greater than or equal to 3 classes of currently marketed antiretroviral agents (NRTIs, NNRTIs, PIs, or fusion inhibitors) at any time prior to screening
* HIV RNA greater than or equal to 5000 copies/mL on a stable ART regimen of at least 3 months of duration
* Greater than or equal to 1 genotypically documented resistance mutation to a reverse transcriptase (RT) inhibitor and greater than or equal to 1 primary resistance mutation to a PI
* Acceptable hematologic, renal, and hepatic laboratory parameters.

Exclusion Criteria:

* No history of recurrent seizure or CNS condition predisposing to seizure
* No active AIDS-defining opportunistic infection
* Subjects who have previously used a CCR5 inhibitor for greater than 4 weeks and/or within 30 days of the screening visit
* Use of any drugs that predispose to seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09-01 (Actual)